CLINICAL TRIAL: NCT04334343
Title: Investigating the Effects of Aerobic and Resistance Training in Vivo on Skeletal Muscle Metabolism in Vitro in Primary Human Muscle Cells (MoTrMyo)
Acronym: MoTrMyo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1436585
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Athletic group (Active Comparator)
  Interventions: Other: Additional Muscle Biopsy Collection
- Sedentary exercise group (Active Comparator)
  Interventions: Other: Additional Muscle Biopsy Collection
- Sedentary no-exercise group (Active Comparator)
  Interventions: Other: Additional Muscle Biopsy Collection

INTERVENTIONS:
Other: Additional Muscle Biopsy Collection — Subjects will be asked if an additional biopsy from an existing incision can be obtained (i.e. additional needle insertion). For each biopsy required in the main MoTrPAC study (NCT03960827), a small needle will be used to inject some numbing medication (similar to what a dentist uses) in your thigh. A small incision (about 1/4 inch) will be made and a special needle will be used to collect 1 or 2 muscle samples (about the size of a pea).

SUMMARY:
The goal of the study is to examine the ability of resistance or aerobic exercise training to "imprint" skeletal muscle cells in a manner which confers long-term changes in this tissue which in-turn contribute to improved metabolic health and functional capacity through epigenetic regulation of novel exercise response genes. This study will also provide primary human skeletal muscle cells to the Molecular Transducers of Physical Activity Consortium (MoTrPAC) (NCT03960827) repository for future use.

ELIGIBILITY:
Inclusion Criteria:

ADULT PARTICIPANT INCLUSION CRITERIA - SEDENTARY PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrPAC Study

  -Willingness to undergo an extra needle insertion for the extra muscle tissue collection during the MoTrPAC muscle biopsy
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged ≥18 y
* Body Mass Index (BMI) >19 to <35 kg/m2
* Sedentary defined as self-reporting no more than 1 day per week, lasting no more than 60 minutes, of regular (structured) EE [e.g., brisk walking, jogging, running, cycling, elliptical, or swimming activity that results in feelings of increased heart rate, rapid breathing, and/or sweating] or RE (resulting in muscular fatigue) in the past year

  * Persons bicycling as a mode of transportation to and from work >1 day/week etc. are not considered sedentary
  * Leisure walkers are included unless they meet the heart rate, breathing, and sweating criteria noted above

ADULT PARTICIPANT INCLUSION CRITERIA - HIGHLY ACTIVE PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrPAC Study

  -Willingness to undergo an extra needle insertion for the extra muscle tissue collection during the MoTrPAC muscle biopsy
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged ≥18 y
* BMI >19 to <35 kg/m2
* Comparator Participants

  * Highly Active Endurance Exercise (HAEE): defined as >240 minutes/week of ET for >1 year; this can include running, walking (brisk, power), cycling, elliptical, etc. which (at a minimum) results in increased heart rate, rapid breathing and sweating
  * Must include cycling at least 2 days/week
  * Highly Active Resistance Exercise (HARE): defined as RT of ≥3 upper and ≥3 lower body muscle groups ≥2 times/week for >1 year; using a prescription sufficient to increase strength and muscle mass
  * Elite or Competitive Athletes: can be included, if they meet HAEE or HARE inclusion criteria
  * Potential participants are informed that use of performance enhancing drugs in the last 6 months is exclusionary
  * In addition to meeting HAEE or HARE inclusion criteria, all HA participants must meet all other exclusion criteria defined in this protocol
  * Individuals who meet inclusion criteria for both HAEE and HARE are exclude

EXCLUSION CRITERIA

ADULT PARTICIPANT EXCLUSION CRITERIA Exclusion criteria are confirmed by either self-report (i.e., medical and medication histories reviewed by a clinician), screening tests performed by the MoTrPAC study team at each clinical site, and/or clinician judgement as specified for each criterion.

* Diabetes (self-report and screening tests)

  * Treatment with any hypoglycemic agents (self-report) or A1c >6.4 (screening test; may reassess once if 6.5-6.7)
  * Fasting glucose >125 (screening test; may reassess once)
  * Use of hypoglycemic drugs (e.g., metformin) for non-diabetic reasons (self-report)
* Abnormal bleeding or coagulopathy (self-report)

  ◦History of a bleeding disorder or clotting abnormality
* Thyroid disease (screening test)

  * Thyroid Stimulating Hormone (TSH) value outside of the normal range for the laboratory
  * Individuals with hypothyroidism may be referred to their primary care provider (PCP) for evaluation and retested; any medication change must be stable for ≥3 months prior to retesting
  * Individuals with hyperthyroidism are excluded, including those with normal TSH on pharmacologic treatment
* Pulmonary (self-report)

  ◦Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Metabolic bone disease (self-report)

  * History of non-traumatic fracture from a standing height or less
  * Current pharmacologic treatment for low bone mass or osteoporosis, other than calcium, vitamin D, or estrogen
* Estrogens, progestins (self-report)

  ◦Supplemental, replacement or therapeutic use of estrogens or progestins within the last 6 months, other than birth control or to control menopausal symptoms
* Pregnancy (screening test) and pregnancy-related conditions (self-report)

  * Pregnant - pregnancy test performed on day of DXA scan in women of child-bearing potential
  * Post-partum during the last 12 months
  * Lactating during the last 12 months
  * Planning to become pregnant during the participation period
* Elevated blood pressure readings (screening test)

  * Aged <60 years: Resting Systolic Blood Pressure (SBP) ≥140 mmHg or Resting Diastolic Blood Pressure (DBP) ≥90 mmHg
  * Aged ≥60 years: Resting SBP ≥150 mmHg or Resting DBP ≥90 mmHg
  * Reassessment of BP during screening will be allowed to ensure rested values are obtained
* Cardiovascular (self-report, screening test, and clinician judgement)

  * Congestive heart failure, coronary artery disease, significant valvular disease, congenital heart disease, serious arrhythmia, stroke, or symptomatic peripheral artery disease (self-report, screening test)
  * Specific criteria used to determine whether a volunteer can undergo the screening Cardiopulmonary Exercise Test (CPET) follow the American Heart Association (AHA) Criteria [54]
  * Inability to complete the CPET
* Abnormal blood lipid profile (screening test)

  * Fasting triglycerides >500 mg/dL
  * Low-density lipoprotein cholesterol (LDL-C) >190mg/dL
* Cancer (self-report)

  * History of cancer treatment (other than non-melanoma skin cancer) and not "cancer-free" for at least 2 years
  * Anti-hormonal therapy (e.g., for breast or prostate cancer) within the last 6 months
* Chronic infection (self-report)

  * Infections requiring chronic antibiotic or anti-viral treatment
  * Human Immunodeficiency Virus
  * Individuals successfully treated for hepatitis C and virologically negative for at least 6 months are not excluded
* Liver enzyme tests (Alanine transaminase, Aspartate transaminase) (screening test)

  ◦>2 times the laboratory upper limit of normal
  * Reassessment during screening may be allowed under some conditions (e.g., recent use of acetaminophen)
  * Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting
* Chronic renal insufficiency (screening test)

  * Estimated glomerular filtration rate <60 mL/min/1.73 m2 from serum creatinine (mg/dL) by the Chronic Kidney Disease Epidemiology Collaboration equation
  * Reassessment may be allowed under some conditions (e.g., questionable hydration status or other acute renal insult)
* Hematocrit (screening test)

  * Hematocrit >3 points outside of the local normal laboratory ranges for women and men
  * Reassessment may be allowed under certain conditions
  * Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting
  * Individuals with known thalassemia trait may be included (despite having >3 points outside of the local normal laboratory ranges), upon approval from their PCP or a hematologist
* Blood donation (self-report)

  * Whole blood donation in the last 3 months or plans for blood donation during the entire protocol period
  * Platelet or plasma donation in the last week or plans for platelet or plasma donation during the entire protocol period
* Autoimmune disorders (self-report)

  ◦Individuals receiving any active treatment (including monoclonal antibodies) within the last 6 months
* Alcohol consumption (self-report)

  * More than 7 drinks per week for women
  * More than 14 drinks per week for men
  * History of binge drinking (≥5 drinks for males or ≥4 drinks for females in a 2-hour period more than once per month)
* Tobacco (self-report)

  ◦Self-reported use ≥3 days/week of tobacco or e-cigarette/e-nicotine products
* Marijuana (self-report)

  ◦Self-reported use ≥3 days/week in any form
* Shift workers (self-report)

  * Night shift work in the last 6 months
  * Planning night shift work during the study period
* Cognitive status (screening)

  ◦Unable to give consent to participate in and safely complete the protocol, as based on the judgement of the local investigator
* Psychiatric illness (self-report and screening test)

  * Hospitalization for any psychiatric condition within one year (self-report)
  * Center for Epidemiological Studies-Depression Scale (CESD) score ≥16 [55] (screening test)
* Weight change (self-report)

  * Weight change (intentional or not) over the last 6 months of >5% of body weight
  * Plan to lose or gain weight during the study
* Lidocaine or other local anesthetic (self-report)

  ◦Known allergy to lidocaine or other local anesthetic
* Other (clinician judgement)

  * Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric or other conditions that, in the opinion of the local clinician, would preclude participation and successful completion of the protocol
  * Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol

EXCLUSIONS FOR MEDICATION USE

* Use of any new drug in the last 3 months
* Dose change for any drug in the last within 3 months
* Cardiovascular

  * Beta blockers and centrally acting anti-hypertensive drugs (clonidine, guanfacine and alpha-methyl-dopa)
  * Anticoagulants (coumadin or Direct Oral Anticoagulants)
  * Antiarrhythmic drugs: amiodarone, dronaderone, profafenone, disopyrimide, quinidine
  * Antiplatelet drugs (other than aspirin ≥100 mg/day): dipyridamole, clopidogrel, ticagrelor
  * Lipid-lowering medications
  * Participants who volunteer to stop lipid-lowering medications for the duration of the study are allowed; inclusion requires lipid-lowering medication to be stopped for 3 months and participant re-evaluated for LDL-C eligibility
* Psychiatric drugs

  * Chronic use of medium or long-acting sedatives and hypnotics (short-acting non-benzodiazepine sedative-hypnotics are allowed)
  * All benzodiazepines
  * Tricyclic antidepressants at a dose ≥75 mg total dose per day
  * Two or more drugs for depression
  * Mood stabilizers
  * Antiepileptic drugs
  * Stimulants, Attention-Deficit/Hyperactivity Disorder (ADHD) drugs
* Muscle relaxants

  ◦Methacarbamol; cyclobenzaprine; tizanidine; baclofen
* Pulmonary, inflammation

  * Chronic oral steroids
  * Burst/taper oral steroids more than once in the last 12 months
  * B2-agonists
  * allowed if on stable dose at least 3 months
* Genitourinary

  * Finasteride or dutasteride
  * Daily phosphodiesterase type 5 inhibitor use
* Hormonal

  * Testosterone, dehydroepiandrosterone, anabolic steroids
  * Anti-estrogens, anti-androgens
  * Growth hormone, insulin like growth factor-I, growth hormone releasing hormone
  * Any drugs used to treat diabetes mellitus or to lower blood glucose
  * Metformin for any indication
  * Any drugs used specifically to induce weight loss
  * Any drugs used specifically to induce muscle growth/hypertrophy or augment exercise-induced muscle hypertrophy
* Pain/inflammation

  * Narcotics and narcotic receptor agonists
  * Regular use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen ≥3 days per week
* Other

  * Anti-malarials
  * Low-potency topical steroids if ≥10% of surface area using rule of 9s
* Any other medications that, in the opinion of local clinicians, would negatively impact or mitigate full participation and completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial function | Week 12 visit
  Tested via a Analysis of Covariance (ANCOVA) with baseline as covariate followed by post-hoc multiple comparisons.
Insulin-stimulated glycogen synthesis in human skeletal muscle cell cultures (HSkMC) | Week 12 visit
  Tested via a Analysis of Covariance (ANCOVA) with baseline as covariate followed by post-hoc multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Sparks, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Kokkinos P, Myers J, Kokkinos JP, Pittaras A, Narayan P, Manolis A, Karasik P, Greenberg M, Papademetriou V, Singh S. Exercise capacity and mortality in black and white men. Circulation. 2008 Feb 5;117(5):614-22. doi: 10.1161/CIRCULATIONAHA.107.734764. Epub 2008 Jan 22. PMID 18212278
- [Background] Egan B, Zierath JR. Exercise metabolism and the molecular regulation of skeletal muscle adaptation. Cell Metab. 2013 Feb 5;17(2):162-84. doi: 10.1016/j.cmet.2012.12.012. PMID 23395166
- [Background] Reaven GM, Chen YD. Role of abnormal free fatty acid metabolism in the development of non-insulin-dependent diabetes mellitus. Am J Med. 1988 Nov 28;85(5A):106-12. doi: 10.1016/0002-9343(88)90402-0. No abstract available. PMID 3057887
- [Background] Snijders T, Nederveen JP, McKay BR, Joanisse S, Verdijk LB, van Loon LJ, Parise G. Satellite cells in human skeletal muscle plasticity. Front Physiol. 2015 Oct 21;6:283. doi: 10.3389/fphys.2015.00283. eCollection 2015. PMID 26557092
- [Background] Ceccarelli G, Benedetti L, Arcari ML, Carubbi C, Galli D. Muscle Stem Cell and Physical Activity: What Point is the Debate at? Open Med (Wars). 2017 Jul 24;12:144-156. doi: 10.1515/med-2017-0022. eCollection 2017. PMID 28765836
- [Background] Murach KA, Fry CS, Kirby TJ, Jackson JR, Lee JD, White SH, Dupont-Versteegden EE, McCarthy JJ, Peterson CA. Starring or Supporting Role? Satellite Cells and Skeletal Muscle Fiber Size Regulation. Physiology (Bethesda). 2018 Jan 1;33(1):26-38. doi: 10.1152/physiol.00019.2017. PMID 29212890
- [Background] Boyle KE, Patinkin ZW, Shapiro ALB, Bader C, Vanderlinden L, Kechris K, Janssen RC, Ford RJ, Smith BK, Steinberg GR, Davidson EJ, Yang IV, Dabelea D, Friedman JE. Maternal obesity alters fatty acid oxidation, AMPK activity, and associated DNA methylation in mesenchymal stem cells from human infants. Mol Metab. 2017 Nov;6(11):1503-1516. doi: 10.1016/j.molmet.2017.08.012. Epub 2017 Sep 1. PMID 29107296
- [Background] Stephens NA, Sparks LM. Resistance to the beneficial effects of exercise in type 2 diabetes: are some individuals programmed to fail? J Clin Endocrinol Metab. 2015 Jan;100(1):43-52. doi: 10.1210/jc.2014-2545. PMID 25412336
- [Background] Ukropcova B, McNeil M, Sereda O, de Jonge L, Xie H, Bray GA, Smith SR. Dynamic changes in fat oxidation in human primary myocytes mirror metabolic characteristics of the donor. J Clin Invest. 2005 Jul;115(7):1934-41. doi: 10.1172/JCI24332. PMID 16007256
- [Background] Aas V, Bakke SS, Feng YZ, Kase ET, Jensen J, Bajpeyi S, Thoresen GH, Rustan AC. Are cultured human myotubes far from home? Cell Tissue Res. 2013 Dec;354(3):671-82. doi: 10.1007/s00441-013-1655-1. Epub 2013 Jun 8. PMID 23749200
- [Background] Berggren JR, Tanner CJ, Houmard JA. Primary cell cultures in the study of human muscle metabolism. Exerc Sport Sci Rev. 2007 Apr;35(2):56-61. doi: 10.1249/JES.0b013e31803eae63. PMID 17417051
- [Background] Gaster M, Kristensen SR, Beck-Nielsen H, Schroder HD. A cellular model system of differentiated human myotubes. APMIS. 2001 Nov;109(11):735-44. doi: 10.1034/j.1600-0463.2001.d01-140.x. PMID 11900052
- [Background] Ciaraldi TP, Abrams L, Nikoulina S, Mudaliar S, Henry RR. Glucose transport in cultured human skeletal muscle cells. Regulation by insulin and glucose in nondiabetic and non-insulin-dependent diabetes mellitus subjects. J Clin Invest. 1995 Dec;96(6):2820-7. doi: 10.1172/JCI118352. PMID 8675652
- [Background] Gaster M. Reduced lipid oxidation in myotubes established from obese and type 2 diabetic subjects. Biochem Biophys Res Commun. 2009 May 15;382(4):766-70. doi: 10.1016/j.bbrc.2009.03.102. Epub 2009 Mar 24. PMID 19324004
- [Background] Lund J, Rustan AC, Lovsletten NG, Mudry JM, Langleite TM, Feng YZ, Stensrud C, Brubak MG, Drevon CA, Birkeland KI, Kolnes KJ, Johansen EI, Tangen DS, Stadheim HK, Gulseth HL, Krook A, Kase ET, Jensen J, Thoresen GH. Exercise in vivo marks human myotubes in vitro: Training-induced increase in lipid metabolism. PLoS One. 2017 Apr 12;12(4):e0175441. doi: 10.1371/journal.pone.0175441. eCollection 2017. PMID 28403174
- [Background] Bourlier V, Saint-Laurent C, Louche K, Badin PM, Thalamas C, de Glisezinski I, Langin D, Sengenes C, Moro C. Enhanced glucose metabolism is preserved in cultured primary myotubes from obese donors in response to exercise training. J Clin Endocrinol Metab. 2013 Sep;98(9):3739-47. doi: 10.1210/jc.2013-1727. Epub 2013 Jul 24. PMID 23884778
- [Background] Consitt LA, Bell JA, Koves TR, Muoio DM, Hulver MW, Haynie KR, Dohm GL, Houmard JA. Peroxisome proliferator-activated receptor-gamma coactivator-1alpha overexpression increases lipid oxidation in myocytes from extremely obese individuals. Diabetes. 2010 Jun;59(6):1407-15. doi: 10.2337/db09-1704. Epub 2010 Mar 3. PMID 20200320
- [Background] Hulver MW, Berggren JR, Carper MJ, Miyazaki M, Ntambi JM, Hoffman EP, Thyfault JP, Stevens R, Dohm GL, Houmard JA, Muoio DM. Elevated stearoyl-CoA desaturase-1 expression in skeletal muscle contributes to abnormal fatty acid partitioning in obese humans. Cell Metab. 2005 Oct;2(4):251-61. doi: 10.1016/j.cmet.2005.09.002. PMID 16213227